CLINICAL TRIAL: NCT06842485
Title: Effectiveness of Telerehabilitation in the Management of Work-Related Musculoskeletal Disorders in Cardiac Sonographers
Brief Title: Effectiveness of Telerehabilitation for Work-Related Musculoskeletal Disorders in Cardiac Sonographers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Shibili Nuhmani, Assistant Porfessor, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-2025-03-0129
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Work Related Musculoskeletal Disorders
Keywords: work related musculoskeletal disorders; cardiac sonographers; tele rehabilitation
MeSH Terms: interventions — Telerehabilitation; Patient Education as Topic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele rehabilitation (Experimental)
- Patient education (Active Comparator)

INTERVENTIONS:
Other: Telerehabilitation — The experimental group will be given a tailored program of telerehabilitation consisting of stretching and strengthening exercises for six weeks (three times per week)
Other: Patient education — Patient education will be given to both the experimental and control groups. Patient education and telerehabilitation will be given to the experimental group. To the control group, patient education alone will be provided

SUMMARY:
Work-related musculoskeletal disorders(WRMDs) are common among cardiac sonographers due to their nature of work. This study aims to find out the effectiveness of the telerehabilitation method in the management of WRMDs among cardiac sonographers. 38 cardiac sonographers diagnosed with WRMDs will be randomly allocated into experimental and control groups with an allocation ratio1:1. The Experimental group will be receiving the telerehabilitation program along with an ergonomic awareness education program for 6 weeks, and the control group will receive an ergonomic awareness education alone. Pain, quality of life and work satisfaction are the outcome measures which will be measured at the baseline and after 6 weeks of the program

ELIGIBILITY:
Inclusion Criteria:

* Cardiac sonographers with work-related musculoskeletal pain.
* Cardiac sonographers practicing adult echocardiography predominantly working in public hospitals, private hospitals or/and private outpatient clinics in Saudi Arabia.

Exclusion Criteria:

* Systematic diseases as reported by the participants such as Diabetes Miletus and Fibromyalgia.
* Using cardiac medications or the pain killer as reported by the participants.
* Any biomechanical abnormalities based on the evaluation of a qualified physical therapist.
* Any other musculoskeletal disorders or injuries which is not related to WRMDs.
* Any recent surgery which may affect the ability to participate in the exercise program.
* Any other contraindications to participate in the exercise program.
* Pregnancy in female participants.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Pain measured by Numeric Pain Rating Scale | baseline and immediately after 6 weeks of the program
  Numeric Pain Rating Scale is a 11-point scale where the minimum score is 0 (indicating no pain) and the maximum score is 10 (representing the worst possible pain)
Quality of life measured by Short Form (36) Health Survey questionnaire | baseline and immediately after 6 weeks of the program
  * The Short Form (36) Health Survey questionnaire contains 36 items that cover eight distinct health domains:
  * Physical Functioning
  * Role Limitations due to Physical Health
  * Role Limitations due to Emotional Problems
  * Energy/Fatigue (Vitality)
  * Emotional Wellbeing (Mental Health)
  * Social Functioning
  * Pain (Bodily Pain)
  * General Health Perceptions
  * Each domain is scored on a scale from 0 to 100.
  * Higher scores indicate better perceived health and quality of life.
Work satisfaction | baseline and immediately after 6 weeks of the program
  Work satisfaction measured by The job satisfaction scale

CONTACTS AND LOCATIONS:
Locations (1):
- Imamabdulrahman bin fasial univeristy, Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes